CLINICAL TRIAL: NCT07029061
Title: Effect of Air Splints on Sensoriomotor Disturbances of the Affected Upper Extremity and Trunk Control in the Adult Post-stroke Patient: A Pilot Randomized Clinical Trial
Brief Title: Effect of Air Splints on Sensoriomotor Disturbances of the Affected Upper Extremity and Trunk Control in the Adult Post-stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alfonso X El Sabio University (Other)
Collaborators: Hospital Beata María Ana (Other)
Responsible Party: Principal Investigator, Alicia Hernando Rosado, Physiotherapist (PhD), Alfonso X El Sabio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universidad Alfonso X El Sabio
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2024-01

CONDITIONS: Stroke Sequelae
Keywords: Physical Therapy; Air splints; Stroke; Upper Limb; Sensorimotor impairments
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application of CPPS (Urias splints) + physiotherapy Intervention Type: Device (Experimental)
  Interventions: Device: Air splints
- Physiotherapy alone following neurodevelopmental approach (No Intervention)

INTERVENTIONS:
Device: Air splints — Application of CPPS (Urias splints) + physiotherapy
  Arms: Application of CPPS (Urias splints) + physiotherapy Intervention Type: Device

SUMMARY:
Objective: Sensory impairment in the affected upper limb occurs in approximately 50% of post-stroke patients and negatively impacts functional capacity and quality of life. This pilot study aims to evaluate whether the standardized use of pneumatic (air) splints, as part of a neurodevelopmental treatment approach, will have a positive effect on sensorimotor deficits in the hemiplegic upper limb of post-stroke patients.

Design: Pilot randomized, single-blind clinical trial.

Setting: Brain injury rehabilitation facility.

Participants: Twenty adults in the subacute phase after stroke will be randomized into two groups. The experimental group (n = 10) will receive air splint therapy combined with physiotherapy (45 minutes per session, twice per week for 4 weeks). The control group (n = 10) will receive only physiotherapy with the same duration and frequency. Sensorimotor outcomes will be assessed using the Fugl-Meyer Assessment for the Upper Extremity (FMA-UE), and finger flexor/extensor strength will be measured using the Amadeo robotic system. Assessments will be conducted before and after the intervention.

Conclusions: The addition of air splints to physiotherapy may enhance exteroceptive and proprioceptive sensitivity in adults recovering from stroke during the subacute phase.

ELIGIBILITY:
Inclusion Criteria:

* Stroke at least 2 months earlier
* Mild/moderate hypertonia (Ashworth ≤3)
* Proprioceptive and exteroceptive deficits
* Trunk stability score between 8-23 (TCT)

Exclusion Criteria:

* Non-vascular etiology
* Clinical instability
* Skin lesions or deformities
* Botulinum toxin in last 3 months
* Cognitive/communication limitations
* Maximum TCT score (23) at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Change in upper limb sensorimotor function measured by the Fugl-Meyer Assessment for the Upper Extremity (FMA-UE) | Baseline and post 4-week intervention
  Change in upper limb sensorimotor function measured by the Fugl-Meyer Assessment for the Upper Extremity (FMA-UE), a validated stroke-specific scale. The FMA-UE ranges from 0 to 66, where higher scores indicate better motor and sensory function.

SECONDARY OUTCOMES:
Change in trunk function measured by the Trunk Control Test (TCT) | Baseline and after 4-week intervention
  Change in trunk function measured by the Trunk Control Test (TCT), which assesses four functional movements. The TCT ranges from 0 to 100, where higher scores indicate better trunk control and functional ability.
Change in balance performance measured by the Mini-Balance Evaluation Systems Test (Mini-BESTest) | Baseline and after 4-week intervention
  Change in balance performance measured by the Mini-Balance Evaluation Systems Test (Mini-BESTest), which ranges from 0 to 28. Higher scores indicate better dynamic balance.
Change in hand strength (flexion and extension) measured using the AMADEO robotic system. | Baseline and after 4-week intervention
  Change in hand strength (flexion and extension) measured using the AMADEO robotic system. Strength will be recorded in Newtons (N). Higher values indicate greater muscle strength.
Change in range of motion (ROM) of the shoulder and fingers measured using the AMADEO robotic system. | Baseline and after 4-week intervention
  Change in range of motion (ROM) of the shoulder and fingers measured using the AMADEO robotic system. ROM will be recorded in degrees (°). Higher values indicate better joint mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Alicia, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No